CLINICAL TRIAL: NCT04186390
Title: Learning Small Bowel Capsule Endoscopy
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anders Bo Nielsen, Medical Doctor, Odense University Hospital
Other Study IDs: OP_736
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Endoscopy; Education; Simulation; Small Bowel Disease; Small Bowel Capsule Endoscopy
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical doctors: Medical doctors with no prior experience in the evaluation of small bowel capsule endoscopy.
  Interventions: Other: Simulation training in small bowel capsule endoscopy

INTERVENTIONS:
Other: Simulation training in small bowel capsule endoscopy — Training in the evaluation of small bowel capsule endoscopies including evaluation, diagnostic and treatment in different cases.

SUMMARY:
This project is a prospective study investigating the education of medical doctors in gastroenterology with no prior experience to evaluate small bowel capsule endoscopies with a diagnostic sensitivity >90%

ELIGIBILITY:
Inclusion Criteria:

* Medical Doctors in medical gastroenterology or surgery

Exclusion Criteria:

* Prior experience with evaluation of small bowel capsule endoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical Doctors in medical gastroenterology or surgery with no prior experience in the evaluation of small bowel capsule endoscopies.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity >90% | 1.5 year
  Percentage of total number of correct diagnostic evaluated cases

SECONDARY OUTCOMES:
Diagnostics | 1.5 year
  Percentage of correct diagnostic description
Clinical consequence | 1.5 year
  Percentage of correct clinical consequence
Total time | 1.5 year
  Total time use for all evaluated cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided